CLINICAL TRIAL: NCT00824369
Title: A Phase 2b Open-Label Rollover Study For Subjects Discontinuing From UK-453,061 Studies For The Treatment Of HIV-1 Infected Subjects
Brief Title: A Rollover Study For Subjects Discontinuing From UK-453,061 Studies For The Treatment Of HIV-1
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer (Industry)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: A5271038
Record Dates: First submitted 2009-01-15; First posted 2009-01-16 (Estimated); Results first posted 2014-08-04 (Estimated); Last update posted 2014-08-04 (Estimated); Status verified 2014-07

CONDITIONS: HIV-1
Keywords: HIV-1; Rollover; Safety.; HIV Infections; treatment experienced
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Anti-retroviral therapy (No Intervention): Anti-retroviral therapy
  Interventions: Drug: No drug will be administered

INTERVENTIONS:
Drug: No drug will be administered — No drug will be administered.

SUMMARY:
The purpose of the protocol is to assess long-term safety and tolerability of subjects who discontinue for any reason from UK-453,061 qualifying studies.

DETAILED DESCRIPTION:
To assess long term safety and tolerability of subjects who discontinue for any reason from UK-453,061 studies. The study will also assess efficacy of the subsequent regimens in these patients. The trial was terminated prematurely on January 29, 2013, due to the decision of the sponsor to discontinue development of lersivirine. The decision to terminate the trial was not based on any safety or efficacy concerns.

ELIGIBILITY:
Inclusion Criteria:

* Previous participation in a qualifying study.
* Male or female at least 18 years of age available for a follow-up period of at least 96 weeks.

Exclusion Criteria:

* Concurrent treatment in another clinical trial.
* Unwilling or unable to be followed for 12 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2009-07; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (25):
- United States (5):
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Dallas, Texas
- Pfizer Investigational Site, Buenos Aires, Argentina
- Brazil (4):
  - Pfizer Investigational Site, Curitiba, Paraná
  - Pfizer Investigational Site, Nova Iguaçu, Rio de Janeiro
  - Pfizer Investigational Site, Campinas, São Paulo
  - Pfizer Investigational Site, São Paulo, São Paulo
- Pfizer Investigational Site, Milan, Italy
- Pfizer Investigational Site, Kota Bharu, Kelantan, Malaysia
- Pfizer Investigational Site, Warsaw, Poland
- Portugal (2):
  - Pfizer Investigational Site, Lisbon
  - Pfizer Investigational Site, Porto
- Puerto Rico (2):
  - Pfizer Investigational Site, Ponce
  - Pfizer Investigational Site, Santurce
- South Africa (2):
  - Pfizer Investigational Site, Dundee, KwaZulu-Natal
  - Pfizer Investigational Site, Cape Town, Western Cape
- Switzerland (2):
  - Pfizer Investigational Site, Lugano
  - Pfizer Investigational Site, Sankt Gallen
- Pfizer Investigational Site, Donetsk, Ukraine
- United Kingdom (3):
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A5271038&StudyName=A%20Rollover%20Study%20For%20Subjects%20Discontinuing%20From%20UK-453%2C061%20Studies%20For%20The%20Treatment%20Of%20HIV-1

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants from two parent studies (A5271015 and A5271022) were included if they discontinued treatment due to virologic failure or other reasons. Participants from 6 countries were enrolled into the A5271015 study and the A5271022 study enrolled participants from 8 countries.
Pre-assignment Details: Twelve and 40 participants who had received: LRV 500 mg QD, LRV 750 mg QD or efavirenz 600 mg QD (in A5271015);or LRV 750 mg QD, LRV 1000 mg QD or etravirine 200 mg BID (in A5271022) were enrolled and treated with open-label antiretrovirals excluding LRV. Data summaries were provided by the randomized treatment groups of the parent protocol.
Groups:
- Participants From A5271015 - Lersivirine 500 mg Arm: Participants who had received lersivirine 500 mg orally once daily in A5271015 parent study
- Participants From A5271015 - Lersivirine 750 mg Arm: Participants who had received lersivirine 750 mg orally once daily in A5271015 parent study
- Participants From A5271015 - Efavirenz 600 mg Arm: Participants who had received efavirenz 600 mg orally once daily in A5271015 parent study
- Participants From A5271022 - Lersivirine 750 mg Arm: Participants who had received lersivirine 750 mg orally once daily in A5271022 parent study
- Participants From A5271022 - Lersivirine 1000 mg Arm: Participants who had received lersivirine 1000 mg orally once daily in A5271022 parent study
- Participants From A5271022 - Etravirine 200 mg Arm: Participants who had received etravirine 200 mg twice daily in A5271022 parent study
Period: Overall Study
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Started | 5 | 4 | 3 | 11 | 12 | 17
Completed | 4 | 4 | 2 | 9 | 11 | 16
Not Completed | 1 | 0 | 1 | 2 | 1 | 1
Not completed — Nolonger willing to participate in study | 1 | 0 | 1 | 2 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm | Total
Number analyzed (Participants) | 5 | 4 | 3 | 11 | 12 | 17 | 52
Age, Customized [Mean (Standard Deviation); unit: years]
  Participants from A5271015 | 33.8 (6.1) | 31.5 (1.7) | 38.3 (3.2) | NA (NA) — This arm belongs to the study A5271022 and not A5271015. | NA (NA) — This arm belongs to the study A5271022 and not A5271015. | NA (NA) — This arm belongs to the study A5271022 and not A5271015. | 34.2 (4.8)
  Participants from A5271022 | NA (NA) — This arm belongs to the study A5271015 and not A5271022. | NA (NA) — This arm belongs to the study A5271015 and not A5271022. | NA (NA) — This arm belongs to the study A5271015 and not A5271022. | 42.7 (9.1) | 39.1 (9.0) | 41.6 (9.4) | 41.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5 | 7 | 11 | 28
  Male | 3 | 2 | 2 | 6 | 5 | 6 | 24

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events, Serious Adverse Events and Participants Who Discontinued Due to Adverse Events
Description: The numbers of participants with treatment emergent adverse events, serious adverse events or discontinuation due to adverse events was reported.
Time Frame: End of Study visit or the Early Termination visit
Population: Safety population consisted of all participants who were enrolled in this study.
Measure: Number; unit: Number of participants
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Number analyzed (Participants) | 5 | 4 | 3 | 11 | 12 | 17
Number of participants
  Number of participants with adverse events | 3 | 4 | 2 | 6 | 7 | 11
  Number of participants with serious adverse events | 0 | 0 | 0 | 0 | 0 | 0
  Participants discontinued due to adverse events | 0 | 0 | 0 | 0 | 0 | 0

2. Secondary Outcome: Number of Participants With Human Immunodeficiency Virus - 1 (HIV 1) Ribonucleic Acid (RNA) Level <50 Copies/mL at Baseline, Month 6, Month 12 and Last Visit
Description: Number of participants with HIV-1 RNA level <50 copies/mL plasma was noted at baseline, month 6, month 12 and last visit.
Time Frame: Baseline, Month 6, Month 12 and Last visit
Population: Analysis population consisted of all participants who were enrolled. The lower limit of quantification of the HIV 1 RNA assays ranged from 20-70 copies/mL as they were performed by local labs. Participants where the HIV-RNA level was with a LLOQ > 50 copies/mL were not included in the analysis at the visit of interest. Only available data was used.
Measure: Number; unit: Number of participants
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Number analyzed (Participants) | 5 | 4 | 3 | 11 | 12 | 17
Number of participants
  Baseline (N = 5, 4, 3, 11, 12, 17) | 2 | 3 | 0 | 9 | 7 | 15
  Month 6 (N = 3, 2, 3, 8, 11, 15) | 2 | 2 | 2 | 5 | 5 | 12
  Month 12 (N = 3, 3, 1, 2, 5, 7) | 2 | 3 | 0 | 2 | 4 | 5
  Last Visit (N = 4, 3, 3, 11, 12, 17) | 3 | 3 | 1 | 7 | 7 | 14

3. Secondary Outcome: Number of Participants With HIV 1 RNA Level <50 Copies/mL or Below the Lower Limit of Quantification (LLOQ) of the Assay at Baseline, Month 6, Month 12 and Last Visit
Description: Number of participants with HIV-1 RNA level <50 copies/mL plasma or below the lower limit of quantification (LLOQ) of the Assay were noted at Baseline, Month 6, Month 12 and Last visit. The lower limit of quantification (LLOQ) of the HIV 1 RNA assays ranged from 20 to 70 copies/mL as the assay was performed by local labs.
Time Frame: Baseline, Month 6, Month 12 and Last visit
Population: Analysis population consisted of all participants who were enrolled in this study. Only available data were used.
Measure: Number; unit: Number of participants
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Number analyzed (Participants) | 5 | 4 | 3 | 11 | 12 | 17
Number of participants
  Baseline (N = 5, 4, 3, 11, 12, 17) | 2 | 3 | 0 | 9 | 7 | 15
  Month 6 (N = 4, 4, 3, 8, 11, 15) | 3 | 4 | 2 | 5 | 5 | 12
  Month 12 (N = 4, 4, 1, 2, 5, 7) | 3 | 4 | 0 | 2 | 4 | 5
  Last Visit (N = 5, 4, 3, 11, 12, 17) | 4 | 4 | 1 | 7 | 7 | 14

4. Secondary Outcome: Absolute Cluster of Differentiation 4+ (CD4+) Cell Count (Cells/uL) at Baseline, Month 6 and Month 12
Description: Participant's immunological status assessed by CD4+ lymphocyte count.
Time Frame: Baseline, Month 6 and Month 12
Population: Analysis population consisted of all participants who were enrolled in this study. Only available data were used.
Measure: Mean (Standard Deviation); unit: cells/uL
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Number analyzed (Participants) | 5 | 4 | 3 | 11 | 12 | 17
cells/uL
  Baseline (N = 4, 4, 3, 11, 12, 17) | 285 (97) | 574 (274) | 564 (121) | 473 (191) | 411 (259) | 455 (212)
  Month 6 (N = 4, 4, 2, 8, 11, 15) | 456 (175) | 514 (195) | 606 (120) | 615 (248) | 413 (266) | 451 (221)
  Month 12 (N = 4, 4, 2, 3, 6, 7) | 618 (285) | 607 (326) | 556 (65) | 378 (57) | 361 (309) | 452 (247)

5. Secondary Outcome: CD4+ Cell Count (Percentage) at Baseline, Month 6 and Month 12
Description: Participant's immunological status assessed by CD4+ lymphocyte count.
Time Frame: Baseline, Month 6 and Month 12
Population: Analysis population consisted of all participants who were enrolled in this study. Only available data were used.
Measure: Mean (Standard Deviation); unit: Percentage of total lymphocytes
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Number analyzed (Participants) | 5 | 4 | 3 | 11 | 12 | 17
Percentage of total lymphocytes
  Baseline (N = 4, 4, 3, 11, 12, 17) | 21 (10) | 29 (9) | 26 (2) | 26 (10) | 21 (12) | 23 (8)
  Month 6 (N = 4, 4, 3, 8, 11, 14) | 36 (14) | 31 (12) | 26 (1) | 28 (12) | 22 (11) | 23 (6)
  Month 12 (N = 4, 4, 3, 3, 6, 6) | 38 (14) | 30 (10) | 27 (7) | 26 (11) | 19 (10) | 18 (7)

ADVERSE EVENTS:
Time Frame: End of Study visit or the Early Termination visit
Description: There were no serious adverse events experienced by the subjects in this study.
Arm/Group | Participants From A5271015 - Lersivirine 500 mg Arm | Participants From A5271015 - Lersivirine 750 mg Arm | Participants From A5271015 - Efavirenz 600 mg Arm | Participants From A5271022 - Lersivirine 750 mg Arm | Participants From A5271022 - Lersivirine 1000 mg Arm | Participants From A5271022 - Etravirine 200 mg Arm
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4 | 0/3 | 0/11 | 0/12 | 0/17
Other Adverse Events (participants affected / at risk) | 3/5 | 4/4 | 2/3 | 6/11 | 7/12 | 11/17
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Participants From A5271015 - Lersivirine 500 mg Arm (N=5) | Participants From A5271015 - Lersivirine 750 mg Arm (N=4) | Participants From A5271015 - Efavirenz 600 mg Arm (N=3) | Participants From A5271022 - Lersivirine 750 mg Arm (N=11) | Participants From A5271022 - Lersivirine 1000 mg Arm (N=12) | Participants From A5271022 - Etravirine 200 mg Arm (N=17)
Abdominal pain lower (Gastrointestinal disorders) | 1 | 3 | 2 | 0 | 0 | 0
Anal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2 | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Varicella (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 1
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Stress (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Epididymitis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1
Cheilitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Frequent bowel movements (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Gastrointestinal disorder (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 1 | 0
Cyst (General disorders) | 0 | 0 | 0 | 0 | 0 | 1
Hepatomegaly (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Seasonal allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Acarodermatitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Onychomycosis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1
Oropharyngeal candidiasis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0
Salpingo-oophoritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 1
Blood glucose increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 1
Blood pressure increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Blood thyroid stimulating hormone increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Low density lipoprotein increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Weight decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 2 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 2
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nerve compression (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1
Breast mass (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.